CLINICAL TRIAL: NCT06450847
Title: Effect of Soleus Muscle Push Ups on Oxidative Stress and Inflammatory Markers, Soleus Endurance, and Adipocytokines Between Type 2 Diabetic, Overweight/Obese and Normal Weight Individuals.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Amenah Hisham Abdelazim, Clinical Instructor, University of Sharjah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USharjah1
Record Dates: First submitted 2024-05-22; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Diabete Type 2; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Active Comparator)
  Interventions: Other: Soleus Muscle Push Up Exercise
- Control group (Placebo Comparator)
  Interventions: Other: Other Exercise

INTERVENTIONS:
Other: Soleus Muscle Push Up Exercise — Members will be asked to do the SPUs for 270 minutes/day for most days of the week (minimum 5 days) for 3 months:
  1. Begin seated on a bench or chair so knees form a 90-degree angle with feet flat on the floor and toes pointed forward. Keep spine straight and shoulders back (not hunched or rounded forward).
  2. Using a slow and controlled tempo, push toes into the floor and lift heels off the ground.
  3. Hold for one to two seconds, pushing down on the balls of feet. Keep your thigh muscles relaxed.
  4. Slowly lower heels and return to start. That's 1 rep. Without shoes Educational session will be given before the intervention time WhatsApp messages will be sent 1-2 times/day to remind the participants to continue doing the exercise and ascertain compliance. Also, the participants are required to daily fill logbook about the duration (in minutes) of the SPU that they did.
  Arms: Interventional group
Other: Other Exercise — Participants will be asked to continue their regular lifestyle
  Arms: Control group

SUMMARY:
The study aims to investigate the impact of Soleus Push Ups (SPU) on Soleus Muscle endurance, Oxidative Stress Markers, Inflammatory markers and Adipocytokines among people in the United Arab Emirates. This will be a pre-post intervention study with participants divided into three groups: Lean normal metabolic profile, metabolically healthy overweight/obese, and patients with Type 2 Diabetes Mellitus. Assessment of anthropometry and body composition, Soleus Muscle Endurance, blood tests for Inflammatory Markers, Oxidative Stress Markers, and Adipocytokines will be conducted pre and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Residents of UAE, both males and females
* Ages 20-50 years
* Uncomplicated Type 2 Diabetic on meds,
* Normal lean BMI
* Overweight and Obese

Exclusion Criteria:

* Recent orthopedic surgery in the LLs
* Pain in the LLs starting from Hips to Ankle.
* Presence of Varicose Veins in the LLs
* Present History of any cardiovascular condition
* Pregnant females
* Morbid Obesity
* Diabetics undergoing Insulin therapy only
* Smokers and alcohol consumption

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Adipocytokine levels in the blood | 3 months
  Measured in μg/ml, using blood test by specialized personnel

SECONDARY OUTCOMES:
Soleus Muscle endurance through Heel Raise Test. • Inflammatory and Oxidative Stress markers through blood sample. | 3 months
  Measured as a number, in repetitions. Detailed procedure described previously.

OTHER OUTCOMES:
BMI | 3 months
  kg/m2
Anthropometric data including weight, height and fat percentage | 3 months
  Measured in kgs, cms and % respectively
Physical Activity and Food habits | 3 months
  Questionnaire (International Physical Activity Questionnaire and Food Frequency Questionnaire)
Venous blood specimens | 3 months
  Measured in mL, using blood test by specialized personnel

IPD SHARING:
Plan to Share IPD: Yes
In case of the need for further expansion of the research, the information might be shared with other researchers in the university without exposure of any personal information or names of participants.